CLINICAL TRIAL: NCT01597050
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Study to Evaluate the Efficacy and Safety of R333 6% Ointment Administered Topically to Discoid Lupus Erythematosus (DLE) and Systemic Lupus Erythematosus (SLE) Patients With Active Cutaneous Discoid Lesions
Brief Title: Safety and Efficacy of Topical R333 in Patients With Discoid Lupus Erythematosus (DLE) and Systemic Lupus Erythematosus (SLE) Lesions
Acronym: SKINDLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C-932333-002
Record Dates: First submitted 2012-05-09; First posted 2012-05-11 (Estimated); Results first posted 2016-06-08 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-06

CONDITIONS: Lupus Erythematosus, Discoid; Lupus Erythematosus, Systemic
Keywords: Discoid Lupus Erythematosus; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Discoid; Lupus Erythematosus, Systemic | interventions — R333

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: R932333 (Active Comparator): R333 6% (60 mg/g), bid
  Interventions: Drug: R932333
- Placebo (Placebo Comparator): Placebo, bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: R932333 — R393233 6% (60 mg/g), bid
  Other Names: R333
  Arms: Drug: R932333
Drug: Placebo — Placebo, bid
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, efficacy and tolerability of topical R333 ointment in Discoid Lupus Erythematosus (DLE) and Systemic Lupus Erythematosus (SLE) patients with active discoid lesions.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled study to evaluate the preliminary efficacy, safety, tolerability, and pharmacokinetics of topical R333 ointment formulated at 6% (60 mg/g) in DLE and SLE patients with active discoid lesions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE or DLE (DLE confirmed histologically prior to randomization).
* At least 2 active discoid lesions secondary to SLE or DLE prior to study entry, each with a minimum Erythema Rating Score of ≥ 2. At least 1 of the active discoid lesions must have been present (by history) for ≥ 3 weeks prior to screening.
* Patients who are taking azathioprine, hydroxychloroquine, chloroquine, quinacrine, methotrexate, and/ or oral glucocorticoids, must be receiving a stable daily dose ≥ 4 weeks prior to randomization and must remain on the same dose throughout the study. Azathioprine, hydroxychloroquine, chloroquine, quinacrine, or methotrexate must be initiated ≥ 8 weeks prior to randomization.

Exclusion Criteria:

* Congenital or acquired immunodeficiency including: HIV infection, agammaglobulinemias, T cell deficiencies or HTLV-1 infection at any time prior to the study.
* Lymphoproliferative disease or previous total lymphoid irradiation.
* Uncontrolled or poorly controlled hypertension.
* History of psoriasis, eczema, or relevant atopy.
* Exposure to excessive or chronic UV radiation (e.g., tanning beds, sunbathing, solarium, phototherapy) within 2 weeks prior to randomization or during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Magilavy, MD, Study Director — Rigel Pharmaceuticals,Inc.
Locations (15):
- United States (12):
  - Wallace Rheumatic Study Center, Los Angeles, California
  - Stanford Dermatology, Redwood City, California
  - Memorial Medical Group Clinical Research Institute, South Bend, Indiana
  - North Shore Long Island Health System, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - University of Pennsylvania-Dermatology Research Office, Philadelphia, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas
  - University of Texas Medical School at Houston, Houston, Texas
  - University of Utah Department of Dermatology, Salt Lake City, Utah
  - Virginia Clinical Research, Inc, Norfolk, Virginia
- Canada (3):
  - University of British Columbia, Vancouver Dermatology Clinical Trials Unit, Vancouver, British Columbia
  - Dermadvances Research, Winnipeg, Manitoba
  - Lynderm Research, Inc, Markham, Ontario

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug: R932333 | Placebo
Started | 36 | 18
Completed | 35 | 18
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: R932333 | Placebo | Total
Number analyzed (Participants) | 36 | 18 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (11.3) | 48.3 (12.57) | 46.8 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 16 | 44
  Male | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 7 | 2 | 9
  United States | 29 | 16 | 45

OUTCOME MEASURES:

1. Primary Outcome: Decrease in the Total Combined Erythema and Scaling Score (Minimum of 0 and Maximum of 65) of All Treated Lesions.
Description: Percentage of patients who achieved at least a 50% decrease from baseline in the total combined Erythema and Scaling score of all treated lesions at Week 4. A decrease is an improvement in measurement of erythema and scaling of the lesions.
Time Frame: Up to Week 4
Population: Per-protocol population all patients who had no major protocol deviations and were present at all scheduled visits up to and including Week 4.
Measure: Number; unit: percentage of subjects
Arm/Group | Drug: R932333 | Placebo
Number analyzed (Participants) | 36 | 18
percentage of subjects | 22.2 | 27.8

ADVERSE EVENTS:
Time Frame: The AE reporting period begins with the first dose of double blind study drug and ends with the final study (follow-up) visit at week 6.
Arm/Group | Drug: R932333 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/18
Other Adverse Events (participants affected / at risk) | 16/36 | 10/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug: R932333 (N=36) | Placebo (N=18)
Upper Respiratory Track Infection (Infections and infestations) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Application site pain (General disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Eyelid margin crusting (Eye disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Application site pruritus (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Mean cell volume increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutrophil count increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
White blood cell count increased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less